CLINICAL TRIAL: NCT06417125
Title: Intranasal Dexmedetomidine Versus Oral Midazolam Premedication for Postoperative Negative Behavior Changes in Children: A Randomized Controlled Trial
Brief Title: Intranasal Dexmedetomidine Versus Oral Midazolam Premedication for Postoperative Negative Behavior Changes in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Collaborators: Fujian Maternity and Child Health Hospital (Other); Fujian Children's Hospital (Unknown)
Responsible Party: Principal Investigator, Yao Yusheng, Clinical Professor, Fujian Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K2024-01-006
Record Dates: First submitted 2024-05-09; First posted 2024-05-16 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Behavior Problem
Keywords: dexmedetomidine; midazolam; postoperative negative behavior change; emergence delirium; tonsillectomy
MeSH Terms: conditions — Mental Disorders; Emergence Delirium | interventions — Dexmedetomidine; Midazolam; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dexmedetomidine group (Experimental): Participants were premedicated with intranasal dexmedetomidine 2 μg/kg and oral sweet solution 0.25 mL/kg.
  Interventions: Drug: Dexmedetomidine Hydrochloride; Drug: Glucose solution
- Midazolam group (Active Comparator): Participants were premedicated with intranasal 0.9% saline 0.02 mL/kg and oral midazolam 0.5 mg/kg.
  Interventions: Drug: Midazolam; Drug: normal Saline
- Placebo group (Placebo Comparator): Participants were premedicated with intranasal 0.9% saline 0.02 mL/kg and oral sweet solution 0.25 mL/kg.
  Interventions: Drug: normal Saline; Drug: Glucose solution

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — Patients were premedicated with intranasal dexmedetomidine 2 μg/kg in the holding area.
  Other Names: Dexmedetomidine hydrochloride Injection
  Arms: Dexmedetomidine group
Drug: Midazolam — Patients were premedicated with oral midazolam 0.5 mg/kg in the holding area.
  Other Names: Midazolam oral solution
  Arms: Midazolam group
Drug: normal Saline — Patients were premedicated with normal saline 0.02 mL/kg in the holding area.
  Arms: Midazolam group; Placebo group
Drug: Glucose solution — Patients were premedicated with oral sweet solution 0.25 mL/kg in the holding area.
  Arms: Dexmedetomidine group; Placebo group

SUMMARY:
The goal of this clinical trial is to learn the effect of dexmedetomidine premedication in postoperative negative behavior changes in children compared to midazolam premedication. It will also learn about the effect of dexmedetomidine and midazolam in emergence delirium. The main questions are:

* Dose dexmedetomidine lower the incidence of postoperative negative behavior changes compared to midazolam?
* Dose dexmedetomidine lower the incidence of emergence delirium compared to midazolam? Researchers will compare dexmedetomidine to midazolam (a common pediatric premedication) to see if dexmedetomidine works to treat postoperative negative behavior change and emergence delirium.

Participants will:

* Take intranasal dexmedetomidine or oral midazolam or placebo (a look-alike substance that contains no drug) premedication
* Fill in the Post hospitalization behavior questionnaire for ambulatory surgery postoperative 1, 3, 7, and 30

DETAILED DESCRIPTION:
Due to the fear of being separated from parents, fear of venipuncture, and facing unfamiliar operating room environment, children have different degrees of anxiety before surgery. Preoperative anxiety can lead to strong stress response and increase the incidence of emergence delirium. It can even cause psychological trauma and affect children's physical and mental health growth. The study showed that preoperative anxiety was positively correlated with the incidence of emergence delirium and postoperative negative behavior change, and emergence delirium was a risk factor for postoperative negative behavior in children.

Currently, midazolam is the most commonly used sedative drug to relieve preoperative anxiety in children. Midazolam has anterograde amnesia effect, reducing the occurrence of intraoperative awareness, and alleviating psychological trauma and memory of malignant stimulation in children. Dexmedetomidine is a highly selective α2 adrenergic agonist with anxiolytic, sedative, and analgesic properties. Our previous study found that preoperative administration of dexmedetomidine can reduce the incidence of emergence delirium in children compared with midazolam However, no clinical studies have directly compared the effects of dexmedetomidine and midazolam premedication on postoperative negative behavior change in children.

This prospective randomized controlled trial was conducted to compare the effects of dexmedetomidine and midazolam premedication on preoperative anxiety, the incidence of postoperative delirium, and postoperative negative behavior changes in children to provide a reference for optimizing clinical anesthesia medication regimens.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I or II;
2. Aged 2-5 years;
3. Scheduled for elective tonsillectomy and (or) adenoidectomy.

Exclusion Criteria:

1. Parents refusing to allow their children to participate;
2. Intake of sedative or analgesic medication within 48 hours before surgery;
3. Developmental delay;
4. Psychosis;
5. Body mass index > 30 kg/m2;
6. Allergy to study drugs;
7. Major life changes 1 month before the operation, such as the divorce of parents, death of parents, moving to a new home, changing to a new kindergarten, etc.;
8. Any other conditions that precluded study inclusion.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 324 (Actual)
Dates: Start 2024-05-22 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative negative behavior changes | Day 7 postoperatively
  Postoperative negative behavior changes will be assessed using the Post Hospitalization Behavior Questionnaire for Ambulatory Surgery (PHBQ-AS).

SECONDARY OUTCOMES:
Incidence of postoperative negative behavior changes | Day 1 postoperatively
  Postoperative negative behavior changes will be assessed using the Post Hospitalization Behavior Questionnaire for Ambulatory Surgery (PHBQ-AS).
Incidence of postoperative negative behavior changes | Day 3 postoperatively
  Postoperative negative behavior changes will be assessed using the Post Hospitalization Behavior Questionnaire for Ambulatory Surgery (PHBQ-AS).
Incidence of postoperative negative behavior changes | Day 30 postoperatively
  Postoperative negative behavior changes will be assessed using the Post Hospitalization Behavior Questionnaire for Ambulatory Surgery (PHBQ-AS).
Incidence of emergence delirium | Within 30 min after extubation
  Emergence delirium will be assessed using the Pediatric Anesthesia Emergence Delirium (PAED) scale (defined as a PAED score of ≥10).
Preoperative anxiety | Before the intervention in holding area
  Preoperative anxiety will be assessed using the modified Yale preoperative anxiety scale. Scores range from 23 to 100 with higher scores indicating greater anxiety.
Length of postanesthesia care unit stay | Up to 60 minutes postoperatively
  Length of postanesthesia care unit stay is defined as the time between arrival in the PACU and readiness for discharge from the PACU (defined as a modified Aldrete score of ≥9).
Emergence time | About up to 30 minutes postoperatively
  Emergence time is defined as the interval from discontinuation of inhalation anesthetic to eye-opening on verbal command.
Parental satisfaction | Postoperative day 1
  Parental satisfaction is self-reported using a five-point Likert scale (5=very satisfied, 4=satisfied, 3=neither satisfied nor dissatisfied, 2=dissatisfied, and 1=very dissatisfied).
Parental separation anxiety | After intervention 30 minutes
  Preoperative sedation level will be measured using the parental separation anxiety scale (PSAS). The PSAS is a 4-point scale as follows: 1=easy separation; 2=whimpers; 3=cries and cannot be easily reassured, but not clinging to parents; and 4=crying and clinging to parents. A PSAS score of 1 or 2 was considered as "acceptable" separation.
Postoperative pain intensity | After extubation 10, 20, 30 min, and postoperative 1 day
  Postoperative pain intensity will be measured using the face, legs, activity, cry, and consolability sacle.
Incidence of adverse events | Up to 24 hours postoperatively
  Adverse events such as bradycardia, tachycardia, hypertension, hypotension, and hypoxia will be recorded during the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochun Zheng, MD, Study Chair — Fujian Provincial Hospital
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
After publication, the individual deidentified participant data underlying published results, the study protocol, and the statistical analysis plan can be accessed upon reasonable request from the corresponding author.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: We would like to share our individual deidentified participant data beginning three months following the publication of the main results.
Access Criteria: All the individual participant data collected during the trial, the study protocol, the statistical analysis plan, and the clinical study report can be accessed with approval from the corresponding author.